CLINICAL TRIAL: NCT04362059
Title: A Clinical Trial of Nebulized Surfactant for the Treatment of Moderate to Severe COVID-19
Acronym: COVSurf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RHM CRI0399
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Patients will be administered surfactant via COVSurf Drug Delivery System
  Interventions: Device: COVSurf Drug Delivery System
- Control Arm (Active Comparator): Patients shall receive regular Standard of Care treatment
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: COVSurf Drug Delivery System — Device introduces surfactant to the patients lungs
  Arms: Treatment Arm
Other: Standard of Care — Standard of care treatment for respiratory illness
  Arms: Control Arm

SUMMARY:
Lung surfactant is present in the lungs. It covers the alveolar surface where it reduces the work of breathing and prevents the lungs from collapsing. In some respiratory diseases and in patients that require ventilation this substance does not function normally. This study will introduce surfactant to the patients lungs via the COVSurf Drug Delivery System

DETAILED DESCRIPTION:
The hypothesis behind the proposed trial of surfactant therapy for COVID-19 infected patients requiring ventilator support is that endogenous surfactant is dysfunctional. This could be due to decreased concentration of surfactant phospholipid and protein, altered surfactant phospholipid composition, surfactant protein proteolysis and/or oedema protein inhibition of surfactant surface tension function and/or oxidative inactivation of surfactant proteins. Variations of these dysfunctional mechanisms have been reported in a range of lung diseases, including cystic fibrosis and severe asthma, and in child and adult patients with ARDS. Our studies of surfactant metabolism in adult ARDS patients showed altered percentage composition of surfactant PC, with decreased DPPC and increased surface tension-inactive unsaturated species, and decreased concentrations of both total PC and phosphatidylglycerol (PG)

The SARS-CoV-2 virus binds to the angiotensin converting enzyme-2 (ACE2) receptor, which is preferentially expressed in the peripheral lung ATII cells. Consequent viral infection of ATII cells could reduce cell number and impair the capacity of the lungs to synthesise and secrete surfactant. This, however, has not yet been demonstrated empirically in COVID-19 patients. If this is the case, then exogenous surfactant administration to the lungs is potential one treatment option to mitigate disease severity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Confirmed COVID-19 positive by PCR
* Within 24 hours of mechanical ventilation (ETI arm) or within 24 hours of needing either CPAP or NIV (CPAP/NIV arm)
* Assent or professional assent obtained

Exclusion Criteria:

* Imminent expected death within 24 hours
* Specific contraindications to surfactant administration (e.g. known allergy, pneumothorax, pulmonary haemorrhage)
* Known or suspected pregnancy
* Stage 4 severe chronic kidney disease or requiring dialysis (i.e., eGFR < 30)
* Liver failure
* Anticipated transfer to another hospital, which is not a study site within 72 hours.
* Current participation or participation in another study within the last month that in the opinion of the investigator would prevent enrollment for safety purposes.
* Consent Declined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Oxygenation Improvement | 3 months
  To assess the improvement in oxygenation as determined by the PaO2/FiO2 ratio after treatment with study treatment
Pulmonary ventilation Improvement | 3 months
  To assess the improvement in pulmonary ventilation as determined by the Ventilation Index (VI), where VI = (Respiratory rate X PIP X PaCo2 (mmHg)/ 1000 after study treatment.
IMV Need | 3 months
  Need for invasive mechanical ventilation (IMV) (CPAP/NIV arm only)

SECONDARY OUTCOMES:
Safety Assessment of Frequency and Severity of Adverse Events | 3 months
  To assess safety as judged by the frequency and severity of adverse events and severe adverse events (SAEs).
Change in PaO2/FiO2 ratio | 3 months
  Mean change in PaO2/FiO2 ratio at 24 and 48 hours after study initiation.
Mean Change in ventilatory index | 48 hours
  Mean change in ventilatory index (VI) at 24 and 48 hours after study initiation
Mean Change in pulmonary compliance | 48 hours
  Mean change in pulmonary compliance (L/cmH2O) at 24 and 48 hours after study initiation in the IMV arm
Mean Change in PEEP requirement | 48 Hours
  Mean change in PEEP (Positive End-Expiratory Pressure) requirement at 24 and 48 hours after study initiation
Clinical Improvement | 28 days
  To evaluate clinical improvement defined by time to one improvement point on an ordinal scale, as described in the WHO master protocol (2020) daily while hospitalised and on days 15 and 28
Mechanical ventilation duration | 3 months
  Duration of mechanical ventilation
Duration of days | 3 months
  Duration of days of IMV or NIV or CPAP
IMV free days | 21 days
  Invasive Mechanical Ventilator (IMV) free days at day 21
Ventilator support free days | 21 days
  Ventilator support (IMV or NIV or CPAP) free days (VSFD) at day 21
Length of ICU stay | 3 months
  Length of intensive care unit stay
Number of days hospitalised | 3 months
  Number of days hospitalised
Mortality | 28 days
  Mortality at day 28

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Grocott, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anzueto A, Baughman RP, Guntupalli KK, Weg JG, Wiedemann HP, Raventos AA, Lemaire F, Long W, Zaccardelli DS, Pattishall EN. Aerosolized surfactant in adults with sepsis-induced acute respiratory distress syndrome. Exosurf Acute Respiratory Distress Syndrome Sepsis Study Group. N Engl J Med. 1996 May 30;334(22):1417-21. doi: 10.1056/NEJM199605303342201. PMID 8618579
- [Result] Surfactant replacement therapy for severe neonatal respiratory distress syndrome: an international randomized clinical trial. Collaborative European Multicenter Study Group. Pediatrics. 1988 Nov;82(5):683-91. PMID 2903480
- [Result] Dushianthan A, Goss V, Cusack R, Grocott MP, Postle AD. Altered molecular specificity of surfactant phosphatidycholine synthesis in patients with acute respiratory distress syndrome. Respir Res. 2014 Nov 7;15(1):128. doi: 10.1186/s12931-014-0128-8. PMID 25378080
- [Result] Goss V, Hunt AN, Postle AD. Regulation of lung surfactant phospholipid synthesis and metabolism. Biochim Biophys Acta. 2013 Feb;1831(2):448-58. doi: 10.1016/j.bbalip.2012.11.009. Epub 2012 Nov 27. PMID 23200861
- [Result] Gunther A, Schmidt R, Harodt J, Schmehl T, Walmrath D, Ruppert C, Grimminger F, Seeger W. Bronchoscopic administration of bovine natural surfactant in ARDS and septic shock: impact on biophysical and biochemical surfactant properties. Eur Respir J. 2002 May;19(5):797-804. doi: 10.1183/09031936.02.00243302. PMID 12030716
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Moller JC, Schaible T, Roll C, Schiffmann JH, Bindl L, Schrod L, Reiss I, Kohl M, Demirakca S, Hentschel R, Paul T, Vierzig A, Groneck P, von Seefeld H, Schumacher H, Gortner L; Surfactant ARDS Study Group. Treatment with bovine surfactant in severe acute respiratory distress syndrome in children: a randomized multicenter study. Intensive Care Med. 2003 Mar;29(3):437-46. doi: 10.1007/s00134-003-1650-1. Epub 2003 Feb 15. PMID 12589529
- [Result] Postle AD, Mander A, Reid KB, Wang JY, Wright SM, Moustaki M, Warner JO. Deficient hydrophilic lung surfactant proteins A and D with normal surfactant phospholipid molecular species in cystic fibrosis. Am J Respir Cell Mol Biol. 1999 Jan;20(1):90-8. doi: 10.1165/ajrcmb.20.1.3253. PMID 9870921
- [Result] Qi F, Qian S, Zhang S, Zhang Z. Single cell RNA sequencing of 13 human tissues identify cell types and receptors of human coronaviruses. Biochem Biophys Res Commun. 2020 May 21;526(1):135-140. doi: 10.1016/j.bbrc.2020.03.044. Epub 2020 Mar 19. PMID 32199615
- [Result] Rebello CM, Jobe AH, Eisele JW, Ikegami M. Alveolar and tissue surfactant pool sizes in humans. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):625-8. doi: 10.1164/ajrccm.154.3.8810596.
- [Result] Rodriguez-Capote K, Manzanares D, Haines T, Possmayer F. Reactive oxygen species inactivation of surfactant involves structural and functional alterations to surfactant proteins SP-B and SP-C. Biophys J. 2006 Apr 15;90(8):2808-21. doi: 10.1529/biophysj.105.073106. Epub 2006 Jan 27. PMID 16443649
- [Result] Schmidt R, Markart P, Ruppert C, Wygrecka M, Kuchenbuch T, Walmrath D, Seeger W, Guenther A. Time-dependent changes in pulmonary surfactant function and composition in acute respiratory distress syndrome due to pneumonia or aspiration. Respir Res. 2007 Jul 27;8(1):55. doi: 10.1186/1465-9921-8-55. PMID 17662121
- [Result] Schwarz KB. Oxidative stress during viral infection: a review. Free Radic Biol Med. 1996;21(5):641-9. doi: 10.1016/0891-5849(96)00131-1. PMID 8891667
- [Result] Shi H, Han X, Jiang N, Cao Y, Alwalid O, Gu J, Fan Y, Zheng C. Radiological findings from 81 patients with COVID-19 pneumonia in Wuhan, China: a descriptive study. Lancet Infect Dis. 2020 Apr;20(4):425-434. doi: 10.1016/S1473-3099(20)30086-4. Epub 2020 Feb 24. PMID 32105637
- [Derived] Dushianthan A, Clark H, Madsen J, Mogg R, Matthews L, Berry L, de la Serna JB, Batchelor J, Brealey D, Hussell T, Porter J, Djukanovic R, Feelisch M, Postle A, Grocott MPW. Nebulised surfactant for the treatment of severe COVID-19 in adults (COV-Surf): A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Dec 10;21(1):1014. doi: 10.1186/s13063-020-04944-5. PMID 33302976
- See also: WHO Master Protocol 2020 — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200301-sitrep-41-covid-19.pdf?sfvrsn=6768306d_2